CLINICAL TRIAL: NCT03594565
Title: The Use of Topical Nasal Steroids for Skin Reactions to Continuous Glucose Monitoring System, Among Children and Youth With Type 1 Diabetes Mellitus: Case Series
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Head of Pediatric Endocrinology Unit, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0277-16-ASF
Record Dates: First submitted 2018-06-17; First posted 2018-07-20 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: T1DM; Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local steroids prior to CGMS insertion (Experimental): topical spraying of fluticasone propionate nasal spray (nsFP) on the skin area of CGMS placement prior to sensor insertion in a group of pediatric T1D patients who had mild to severe local skin reactions to CGMS adhesives.
  Dosage: 2 puffs.
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Local Fluticasone Propionate use prior to continuous glucose monitoring system insertion

SUMMARY:
Background Type 1 diabetes mellitus is a chronic metabolic disorder that presents a significant set of challenges to the patient, their family and the physician. Near normoglycemia is associated with a reduced risk of microvascular and macrovascular complications in type 1 diabetes mellitus but is difficult to achieve despite considerable effort from patients and healthcare providers . Furthermore, episodes of hypoglycemia are frequent and may endanger life acutely. Subcutaneous glucose monitoring systems (CGMS), also called sensors that continuously measure interstitial fluid glucose levels have become available recently, and approved for use in children. CGMS has made it possible to assess the patterns and trends of blood glucose and the substantial variability in glucose excursions in the population of type 1 diabetes, and to prevent severe hypoglycemic episodes. The benefits of this technology are most apparent with near continuous wear of the sensors and is incorporated into the day to day management of the individual's diabetes . These devices provide patients with information regarding postprandial and overnight glucose profiles that are rarely, if ever, obtained with conventional self monitoring of blood glucose using home glucose meters .

Skin reactions CGM systems measure the glucose content of interstitial fluid , using an electrochemical enzymatic sensor, which is accessed by a needle sensor inserted subcutaneously. The CGMS is compromised of a disposable subcutaneous glucose-sensing catheter connected by a cable to a pager sized glucose monitor . Problems related associated to skin irritation and sensor adhesiveness in these young children presents challenges to daily use of the CGMS. In the study conducted by Englert et al, for the Diabetes Research in Children (Directnet) Study Group - three primary factors that contributed to reduced CGM use were identified: the limited body surface area in smaller children, ambient temperature and humidity, as well as the type and duration of physical activity. A study conducted in Israel, by our group, demonstrated only 30% consistant use of the system, partly due to skin reactions . In our cohort, thirty participants of the CGMS group (36.1 %) had signs of local reaction to the RT-CGMS insertion. Mild-to severe local redness was reported in 19 % of patients and hyperpigmentation in 17 %. Skin reactions were among the reasons for discontinuation of CGMS (2/51 participants, 3.9 %).

The use of Local Fluticasone for dermatological use Fluticasone propionate - the first carbothioate corticosteroid - has been classified as a potent anti-inflammatory drug for dermatological use. It is available as cream and ointment formulations for the acute and maintenance treatment of patients with dermatological disorders such as atopic dermatitis, psoriasis and vitiligo. This glucocorticoid is characterized by high lipophilicity, high glucocorticoid receptor binding and activation, and a rapid metabolic turnover in skin. Several clinical trials demonstrate a low potential for cutaneous and systemic side-effects . Even among paediatric patients with atopic dermatitis, fluticasone propionate proved to be safe and effective. These pharmacological and clinical properties are reflected by the high therapeutic index of this glucocorticoid. The same drug is also available as a nasal spray ,for cases of allergic rhinitis.

The use of fluticasone in spray, sprayed on the location of CGMS insertion, prior to insertion to prevent adverse skin reactions in patients with type 1 DM using CGMS devices has not been addressed in the literature.

Hypothesis :

Minimizing skin irritation may significantly improve duration of use and tolerability of CGM devices by young children, as well a in young adults. The Investigators assumed that the simple use of a spray, which will not decrease the adhesiveness of the sensor, may improve use .

Methods Children whose parents had difficulty with CGMS due to irritation, redness were offered to use Flixonase (FLUTICASONE PROPIONATE), with an approval form 29ג, indicating it is not approved for this specific diagnosis .

The investigators followed those patients for improvement and possible local side effects.

Study population Every patient, treated by the pediatric and adolescents diabetes mellitus interdisciplinary service , Assaf Haroffe Medical Center , who experienced local reaction at the site of CGMS was offered this medical option .

Charts were reviewed for response . total participants - 15

ELIGIBILITY:
Inclusion Criteria:

* Age 1-20 years
* Local skin reaction to CGMS indicating local or systemic management.

Exclusion Criteria:

* Patients who were offered nsFP but did not actually use it.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Difference in skin irritation before and after regular application of nsFP according to the modified Draize scale. | 2 years from patient first enrollment
  Erythema and edema were assessed for adhesive and sensor-insertion areas on a 4-point scale, with total score ≤3 defined as mild, 4-5 as moderate, and 6-8 as severe.

SECONDARY OUTCOMES:
Change in BMI SDS | 6 months after nsFP use
  Weight (kg), height (meters), age (years) and sex will be combined to report BMI SDS
Change in height SDS 6 months after nsFP use | 6 months after nsFP use.
  Height (meters), age (years) and sex will be combined to report height SDS
Change in mean glucose 6 months after nsFP use | 6 months after nsFP use.
  Mean glucose measured as mg/dl
Change in glycated hemoglobin 6 months after nsFP use | 6 months after nsFP use.
  Glycated hemoglobin measured with the DCCT (Diabetes Control and Complications Trial) units, presented as percentage
  The new mmols/mol values are known as the IFCC (International Federation of Clinical Chemistry) units.

IPD SHARING:
Plan to Share IPD: Undecided